CLINICAL TRIAL: NCT03267056
Title: Real-World Registry Assessing the Clinical Use of the Orchid Drug Coated Balloon Catheter
Brief Title: AcoArt IV / SFA in China:Drug-eluting Balloon for SFA Angioplasty Evaluation in China
Status: Completed | Type: Observational
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Acotec-04
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-04

CONDITIONS: Peripheral Artery Disease
Keywords: drug-coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCB arm: drug eluting balloon catheter
  Interventions: Device: drug eluting balloon catheter (trade name: Orchid)

INTERVENTIONS:
Device: drug eluting balloon catheter (trade name: Orchid) — use drug eluting balloon catheter(trade name: Orchid) to inflate the stenosis or occlusion in superficial femoral artery(SFA) and/or popliteal artery

SUMMARY:
The registry is a prospective, multicenter, single arm post-market real-world registry in China assessing the clinical use, safety and outcomes of the Orchid 035 DCB Catheter in the Superficial Femoral Artery (SFA) and Popliteal Arteries (PA).

DETAILED DESCRIPTION:
PTA is an established alternative to open surgical bypass for the treatment of infrainginual disease of critical limb ischemia.

DEBs are designed to promote arterial patency by reducing neointimal proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients with peripheral artery disease (PAD), with Rutherford classification between 2 and 5
* an occlusion or a minimum grade of stenosisPrimary over 70% in the superficial femoral artery an /or the popliteal artery
* Total length of treat lesion(s)is less or equal to 20cm
* signed Patient informed consent form

Exclusion Criteria:

* plasma Cr level greater than 150 umol/L in patients
* patients with acute thrombosis requiring lysis or thrombectomy
* 2 or more than 2 stenosis lesions in traget vessel
* patient with a lysis or an lower limb intervention as a therapy within the last 6 weeks
* patient requiring intervention in both lower limbs at the same time
* have >30% residual stenosis or blood-limited dissection after predilation
* distal outflow through less than one lower leg vessel
* known hypersensitivity to aspirin, heparin, clopidogrel,paclitaxel, contrast medium, etc.
* patients participating in another clinical trials with interfere with this trial in the past 3 months
* pregnancy and lactating woman
* untreatable bleeding diatheses
* other diseases, such as cancer, liver disease, or cardiac insufficiency, which may lead to protocol violations or markedly shorten a patients's life expectancy(less than 1 years)
* patients unable or unwilling to participate this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a more than 70% stenosis at femoral and/or popliteal artery meet all the inclusion and excluison criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Primary patency of target lesion. | 12 months
  The primary efficacy end point was primary patency at 12 months following the index procedure, defined as freedom from clinically driven target lesion revascularization and restenosis as determined by a duplex ultrasonography-derived peak systolic velocity ratio of
  ≤2.4

SECONDARY OUTCOMES:
target lesion revascularization,target lesion revascularization is defined as any reintervention of artery bypass graft surgery involving the target lesion | 6 months, 12 months
  target lesion revascularization is defined as any reintervention of artery bypass graft surgery involving the target lesion
improvment in Rutherford stage | 6 months, 12 months
  improvementin Rutherford stage is defined as an upward shift of at least 1 category on Rutherford classification as compared to baseline
change in ankle brachial index(ABI) | 12 months
  change in ankle brachial index(ABI) compared to baseline
Device success during the operation | during the operation
  Device success is defined as successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below the rated burst pressure (RBP).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Chinese PLA General Hospital; Yinghua Zou, Principal Investigator — Peking University First Hospital
Locations (10):
- China (10):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The second hospital of hebei medical university, Shijiazhuang, Hebei
  - The second affiliated hospital of Harbin medical university, Harbin, Heilongjiang
  - Wuhan central hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Tianjin First Center Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Nanjing, Zhejiang